CLINICAL TRIAL: NCT05878899
Title: Postpartum Heparin Against Venous Thromboembolism: a Pilot Randomized Controlled Trial
Acronym: PP-HEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Blondon, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UGeneva 2021-02350
Record Dates: First submitted 2023-03-06; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxaparin (Experimental): Enoxaparin 20-60mg o.d., according to bodyweight, for 10 days postpartum.
  Interventions: Drug: Enoxaparin
- No treatment (No Intervention): No treatment.

INTERVENTIONS:
Drug: Enoxaparin — Prophylactic dose of enoxaparin once daily for 10 days after delivery.
  Arms: Enoxaparin

SUMMARY:
In previous attemps to answer the question of risk-benefit of postpartum thromboprophylaxis, researchers were faced with low recruitement rates. The goal of this pilot feasibility randomized controlled trial of postpartum pharmacological thromboprophylaxis is to examine the feasibility (recruitement rate) and participation rate at the Geneva University Hospitals

ELIGIBILITY:
Inclusion Criteria: adult women within 48h of delivery, with:

* ≥2 of the following risk factors Age ≥35 years Pre-pregnancy BMI 30.0-34.9kg/m2 Current smoking Elective cesarean section Postpartum hemorrhage Antenatal immobility
* and/or ≥1 of the following risk factors: Emergency cesarean section Pre-pregnancy BMI ≥35kg/m2 Known low-risk thrombophilia (heterozygous factor V Leiden; heterozygous G20210 prothrombin mutation) Pre-eclampsia Pre-term delivery (<37th week of gestation) Peripartum systemic infection (defined as fever with use of antibiotics) Intra-uterine growth restriction (birth weight <5th percentile)

Exclusion Criteria:

* any indication for therapeutic anticoagulation
* a high-risk of postpartum venous thromboembolism (personal history, high-risk thrombophilia)
* an increased bleeding risk
* a contra-indication to the use of heparin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Recruitement rate | 6 months
  Number of study inclusion per month
Study participation | Within 48 hours after delivery
  Proportion of eligible women who are presented the study and who accept to participate

SECONDARY OUTCOMES:
Venous thromboembolism | Within 90 day after delivery
  Pulmonary embolism and deep vein thrombosis
Bleeding | Within 90 day after delivery
  Major and clinically relevant non-major bleeding
Surgical site complication | Within 90 day of delivery
  Cesarean section site complication
Heparin-induced thrombocytopenia | Within 90 day of delivery
Septic pelvic thrombophlebitis | Within 90 day of delivery
All-cause mortality | Within 90 day of delivery
Satisfaction with study intervention | After completion of the 10 days of study drug
  Satisfaction based on TSQMII questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blondon M, Claver M, Celetta E, Righini M, de Tejada BM. Preventing Postpartum Venous Thromboembolism With Low-Molecular-Weight Heparin: The PP-HEP Pilot Randomised Controlled Trial. BJOG. 2025 Jan;132(1):35-43. doi: 10.1111/1471-0528.17943. Epub 2024 Sep 5. PMID 39238110